CLINICAL TRIAL: NCT01757561
Title: The Difference in Cerebral Oxygenation Between Propofol and Sevoflurane
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun-ying Guo, Attending physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 伦审[2012]324号
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Cerebral Hypoxia; Postoperative Cognitive Dysfunction
Keywords: jugular bulb oxygen saturation; postoperative cognitive dysfunction; propofol; sevoflurane
MeSH Terms: conditions — Hypoxia, Brain; Postoperative Cognitive Complications | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Propofol-Abnormal: patients with preoperative SjvO2<55%,using the TIVA technology with propofol,
  Interventions: Procedure: propofol
- Propofol-Normal: patients with preoperative SjvO2≥55%,using the TIVA technology with propofol,
  Interventions: Procedure: propofol
- Sevoflurane-Abnormal: patients with preoperative SjvO2<55%,using the VIMA technology with sevoflurane,
  Interventions: Procedure: sevoflurane
- Sevoflurane-Normal: patients with preoperative SjvO2≥55%,using the VIMA technology with sevoflurane,
  Interventions: Procedure: sevoflurane

INTERVENTIONS:
Procedure: propofol — use total intravenous anesthesia with propofol
  Groups: Propofol-Abnormal; Propofol-Normal
Procedure: sevoflurane — use inhalation anesthesia with sevoflurane
  Groups: Sevoflurane-Abnormal; Sevoflurane-Normal

SUMMARY:
the purpose of this study is to investigate whether propofol and sevoflurane have difference effect on cerebral oxygenation .

DETAILED DESCRIPTION:
the purpose of this study:(1) to investigate the incidence of preoperative cerebral oxygenation abnormity (SjvO2 <55%) and its relationship with intraoperative cerebral desaturation and POCD. (2) To investigate the change of intraoperative cerebral oxygen supply and demand balance and the incidence of cerebral desaturation in patients with abnormal preoperative cerebral oxygenation during sevoflurane anesthesia. (3)To investigate the incidence of early POCD in patients with abnormal preoperative cerebral oxygenation during sevoflurane and propofol anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to take major surgery under general anesthesia over 18 years old classified as ASA class three or less

Exclusion Criteria:

* have a diagnosis of cerebrovascular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective major surgery
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guo J Ying, Master, Study Chair — the First Affiliated Hospital of SunYetSen University
Locations (1):
- the First Affiliated Hospital of Sun YetSen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol-Abnormal: patients with preoperative SjvO2<55%
  propofol: use total intravenous anesthesia with propofol
- Propofol-Normal: patients with preoperative SjvO2≥55%
  propofol: use total intravenous anesthesia with propofol
- Sevoflurane-Abnormal: patients with preoperative SjvO2<55%
  sevoflurane: use inhalation anesthesia with sevoflurane
- Sevoflurane-Normal: patients with preoperative SjvO2≥55%
  sevoflurane: use inhalation anesthesia with sevoflurane
Period: Overall Study
Arm/Group | Propofol-Abnormal | Propofol-Normal | Sevoflurane-Abnormal | Sevoflurane-Normal
Started | 38 | 34 | 38 | 34
Completed | 32 | 28 | 31 | 25
Not Completed | 6 | 6 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol-Abnormal | Propofol-Normal | Sevoflurane-Abnormal | Sevoflurane-Normal | Total
Number analyzed (Participants) | 32 | 28 | 31 | 25 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (7.6) | 69 (10.5) | 64.2 (8.3) | 67.2 (8.5) | 65.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 8 | 8 | 38
  Male | 23 | 15 | 23 | 17 | 78
ASA [Number; unit: participants] — ASA I No organic, physiologic, biochemical or psychiatric disturbance ASA II A patient with mild systemic disease that results in no functional limitation. Examples: well-controlled hypertension, uncomplicated diabetes mellitus.
  ASA III A patient with severe systemic disease that results in functional impairment ASA IV Severe systemic disease that is a constant threat to life. ASA V Moribund condition in a patient who is not expected to survive with or without the operation.
  ASA VI Declared brain death patient whose organs are being harvested for transplantation.
  participants
    ASAⅡ | 30 | 22 | 23 | 17 | 92
    ASA Ⅲ | 2 | 6 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Intraoperative Desaturation Between Propofol and Sevoflurane General Anesthesia
Description: SjvO2 were measured before anesthesia, after intubation, every hour during operation, after extubation by jugular vein blood and atrial blood gas analysis.The incidence of intraoperative cerebral desaturation was recorded when SjvO2<50%.
Time Frame: baseline ,every hour in the operation period,after extubation
Measure: Number; unit: participants
Arm/Group | Propofol-Abnormal | Propofol-Normal | Sevoflurane-Abnormal | Sevoflurane-Normal
Number analyzed (Participants) | 32 | 28 | 31 | 25
participants | 17 | 6 | 6 | 0

2. Secondary Outcome: the Incidence of Postoperative Cognitive Disfunction(POCD)Between Propofol and Sevoflurane General Anesthesia
Description: The incidence of early POCD was recorded. The MMSE score and the Montreal cognitive assessment (MoCA) score were recorded 1day before surgery, 1-3 day after surgery and 5-7 day after surgery. The POCD was defined as MMSE score illiterate group ≤ 17, primary and secondary school group ≤ 20, junior high school and above group ≤ 24，or the MoCA score decreased 20% with the baseline.
Time Frame: 1-3days、5-7days after operation
Measure: Number; unit: participants
Arm/Group | Propofol-Abnormal | Propofol-Normal | Sevoflurane-Abnormal | Sevoflurane-Normal
Number analyzed (Participants) | 32 | 28 | 31 | 25
participants
  1--3days after operation | 9 | 4 | 4 | 8
  5-7 days after operation | 5 | 2 | 4 | 4

3. Secondary Outcome: the Change in the Level of Serum BDNF(Brain-derived Neurotrophic Factor ) Between Propofol and Sevoflurane Anesthesia
Time Frame: before anesthesia, after extubation ,1day after operation
Reporting Status: Not Posted

4. Secondary Outcome: the Change in the Level of Serum s-100β Between Propofol and Sevoflurane Anesthesia
Time Frame: before anesthesia,after extubation,1 day after operation
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Vital Signs
Description: heart rate, artery blood pressure,pulse oxygen saturation,temperature
Time Frame: baseline , evey hour in the operation,afte extubation
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Blood Gas Analysis
Description: including artery blood and blood from jugular vein bulb
Time Frame: baseline,every hour in the operation,after extubation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: the day of surgery and 1 week after surgery
Arm/Group | Propofol-Abnormal | Propofol-Normal | Sevoflurane-Abnormal | Sevoflurane-Normal
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/34 | 0/38 | 0/34
Other Adverse Events (participants affected / at risk) | 1/38 | 0/34 | 0/38 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol-Abnormal (N=38) | Propofol-Normal (N=34) | Sevoflurane-Abnormal (N=38) | Sevoflurane-Normal (N=34)
heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol-Abnormal (N=38) | Propofol-Normal (N=34) | Sevoflurane-Abnormal (N=38) | Sevoflurane-Normal (N=34)
allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes